CLINICAL TRIAL: NCT06986798
Title: Exploratory Study to Investigate the Association Between the Onset of Disseminated Intravascular Coagulation (DIC) and Disease Progression With Different Biomarker Candidates as Well as Standard Clinical and Demographic Parameters in Adult Patients With Sepsis
Brief Title: A Study to Learn About the Occurrence of Disseminated Intravascular Coagulation in People With Sepsis and Further Worsening of Sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 22795
Record Dates: First submitted 2025-04-24; First posted 2025-05-23 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Sepsis; Sepsis Associated DIC
Keywords: Sepsis; DIC
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Septic participants in ICU (Other): The study population will consist of septic participants admitted to a medical intensive care unit (ICU), as defined in the inclusion criteria. No investigational study interventions will be administered in this study. Participants will undergo therapeutic and diagnostic procedures as per local standard medical care and as deemed appropriate by the treating physicians. Collection of blood and of available clinical data are the only activities performed in addition.
  Interventions: Other: Local standard medical care

INTERVENTIONS:
Other: Local standard medical care — No investigational study interventions will be administered in this study. Participants will undergo therapeutic and diagnostic procedures as per local standard medical care and as deemed appropriate by the treating physicians. Collection of blood and of available clinical data are the only activities performed in addition.

SUMMARY:
This is an exploratory study in which data from people with sepsis (a serious condition in which the body responds to an infection that damages vital organs) admitted to an Intensive care unit (ICU) who will receive treatment are studied.

Sepsis is a serious condition that happens when the body's reaction to an infection causes organ damage. Disseminated intravascular coagulation (DIC) is a serious blood disorder that can cause clots throughout the body, blocking blood vessels. DIC is a serious condition that can happen in people with sepsis, which may further lead to organ damage or even death.

No investigational products will be administered in this study. Participants will be treated with the standard of care (SOC) for sepsis. The SOC is the treatment that medical experts consider most appropriate currently.

There are limited treatments available for DIC, especially for people with sepsis and other diseases. To better understand the impact of sepsis, and how it develops into DIC, more knowledge is needed in the European population.

The main purpose of this study is to learn about how sepsis worsens, especially from the time a person is admitted to the ICU until they develop DIC. To do this, researchers will identify certain biomarkers to understand how DIC develops and progresses in people with sepsis. A biomarker is present in blood, other body fluids, or tissues and indicates a disease or abnormal process inside the body.

To learn about this, researchers will collect information about the participants who develop DIC, including cause, and severity of DIC (using a score called ISTH DIC Score). The data will be collected from participants' hospital records in more than three European countries. Each participant will be in the study for up to 56 days. During the study, the doctors and their study team will take blood samples up to 6 times to check for the presence of biomarkers for the identification of people with DIC.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 years of age inclusive, at the time of signing the informed consent.
* Participants with diagnosed sepsis according to sepsis-3 definition.
* Participants with documented suspected origin of infection.
* Informed consent of capable participant or, in case of participant being incapable of giving informed consent, consent for study inclusion will be sought according to applicable laws and regulations.

Exclusion Criteria:

* Patients deferred from other Intensive Care Units (ICUs).
* Patients longer than 24 hours on ICU.
* Known coagulation disorder.
* Ongoing active clinically significant bleeding.
* Participants experienced trauma or major surgery (within 4 weeks).
* Active malignancy.
* Decompensated liver impairment Child-Pugh Class C.
* Moribund patients not expected to survive 24 hours (clinical decision).
* Ongoing therapeutic anticoagulation (prophylactic dose of Unfractionated Heparin [UFH]/Low Molecular Weight Heparin [LMWH] is allowed) or antiplatelet therapy (except low dose [≤100 mg] acetyl salicylic acid [ASA]). If previously named treatment can be stopped the participants will be eligible if a "wash out"-time of five half-lives is applied before start of study.
* Patients who have received any investigational drug involving pharmacological interventions, or biological or cell therapy interventions or prohibited therapy within 28 days or five half-lives, whichever is longer, prior to screening/baseline.
* Any reason that would make participation unadvisable, at the discretion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2025-01-29 (Actual); Primary Completion 2025-12-22 (Actual); Study Completion 2026-02-02 (Actual)

PRIMARY OUTCOMES:
Occurrence of Disseminated Intravascular Coagulation (DIC) as defined by ISTH criteria | Until Day 56
  The International Society on Thrombosis and Haemostasis (ISTH) developed a scoring system to aid in the diagnosis and management of DIC. The ISTH DIC score is a standardized tool that quantifies the severity of DIC based on specific laboratory parameters. The total score ranges from 0 to 8, with a score of ≥ 4 indicating overt DIC. In this study, the ISTH DIC score will be employed for screening purposes as well as to evaluate the presence and severity of DIC in participants enrolled.

SECONDARY OUTCOMES:
Sequential Organ Failure Assessment (SOFA) score at baseline | At baseline
  The Sequential Organ Failure Assessment (SOFA) score is a clinical tool used to track a patient's status in regard to the organ systems during stay in an Intensive Care Unit (ICU), assigning a score from 0 (normal function) to 4 (high degree of dysfunction) for each system. The total SOFA can range from 0 to 24.
Change from baseline in SOFA score on Day 5 or End of ICU stay, whichever happens first | Baseline and Day 5 or End of ICU stay
  The Sequential Organ Failure Assessment (SOFA) score is a clinical tool used to track a patient's status in regard to the organ systems during stay in an Intensive Care Unit (ICU), assigning a score from 0 (normal function) to 4 (high degree of dysfunction) for each system. The total SOFA can range from 0 to 24.
All-cause mortality until Day 56 | Until Day 56
Type of organ support status until Day 56 | Until Day 56
  Describe the type of organ support status.
Time with organ support status until Day 56 | Until Day 56
  Describe the time with organ support status.
Type of hospitalization status until Day 56 | Until Day 56
  Describe the type of hospitalization (ICU [Intensive Care Unit]/ common ward/ discharge).
Time with hospitalization until Day 56 | Until Day 56
  Describe the time with hospitalization.

CONTACTS AND LOCATIONS:
Locations (31):
- Austria (3):
  - MedUni Innsbruck | Innere Medizin I, Internistische Intensiv- und Notfallmedizin, Innsbruck, Tyrol
  - MedUni Graz | Innere Medizin, ICU, Graz
  - MedUni Wien | Univ. Klinik für Klinische Pharmakologie, Vienna
- Belgium (4):
  - AZ Groeninge - Campus Kennedylaan, Kortrijk
  - Centre Hospitalier Universitaire (CHU) de Liege - Domaine Universitaire du Sart Tilman, Liège
  - Clinique Saint-Pierre d'Ottignies - Intensive Care, Ottignies-Louvain-la-Neuve
  - Universite Catholique de Louvain (UCL) - Cliniques Universitaires Saint-Luc, Woluwe-Saint-Lambert
- France (7):
  - Centre Hospitalier Universitaire d'Angers - Médecine Intensive Réanimation et Médecine Hyperbare, Angers
  - Hôpital Raymond-Poincaré - Service de Médecine Intensive - Réanimation, Médecine Hyperbare, Garches
  - Centre Hospitalier Départemental Vendée - Service de réanimation polyvalente, La Roche-sur-Yon
  - Centre Hospitalier Universitaire de Limoges Dupuytren 1 - Service de réanimation polyvalente, Limoges
  - Hopital Hotel Dieu Nantes - Service de Médecine Intensive Réanimation, Nantes
  - Hopitaux Universitaires de Strasbourg Nouvel Hopital Civil - Service de Médecine Intensive Réanimation, Strasbourg
  - CHRU de Tours - Hôpital Bretonneau - Médecine Intensive Réanimation, Tours
- Germany (5):
  - Kliniken der Stadt Köln gGmbH - Krankenhaus Merheim - Lungenklinik, Cologne, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus an der Technischen Universitaet Dresden | Medizinische Klinik I - FB Haemostaseologie, Dresden
  - Universitaetsklinikum Essen | Klinik für Anaesthesiologie und Intensivmedizin, Essen
  - RKH Klinikum Ludwigsburg, Ludwigsburg
  - Klinikum der Universität München AöR - Klinik für Anaesthesiologie (Campus Großhadern), München
- Italy (4):
  - Azienda Ospedaliero-Universitaria Di Bologna IRCCS_Policlinico Sant'Orsola - Anestesia e TI Polivalente, Bologna
  - Azienda Socio Sanitaria Territoriale Santi Paolo e Carlo_Ospedale S. Carlo - Anestesia e Rianimazione, Milan
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Anestesia, Rianimazione, Terapia Intensiva e Tossicologia Clinica, Roma
  - Humanitas Mirasole S.p.A. - Anestesia e Terapie Intensive, Rozzano
- Netherlands (3):
  - Medisch Spectrum Twente - Intensive Care, Enschede
  - Universitair Medisch Centrum St. Radboud, Nijmegen
  - Maasstad, Rotterdam
- Spain (5):
  - Hospital Universitario De Getafe | Unidad de Cuidados Intensivos, Getafe, Madrid
  - Hospital Universitario Central De Asturias | Unidad de Cuidados Intensivos, Oviedo, Principality of Asturias
  - Hospital Universitari Vall D Hebron | Unidad de Cuidados Intensivos, Barcelona
  - Hospital Clinico San Carlos | Unidad de Cuidados Intensivos, Madrid
  - Hospital Universitario Virgen Del Rocio S.L. | Unidad de Cuidados Intensivos, Seville

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.